CLINICAL TRIAL: NCT05271136
Title: A Double-blind, Randomized, Controlled Clinical Study to Evaluate the Efficacy of an Anti-Aging Serum
Brief Title: A Clinical Study to Evaluate the Efficacy of an Anti-Aging Serum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Collaborators: Stephens & Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C20-D146
Record Dates: First submitted 2021-09-29; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Fine Lines; Wrinkle; Photoaging
Keywords: anti-aging; serum
MeSH Terms: interventions — cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion; Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, controlled, single-center
Who Masked: Participant, Investigator
Masking Description: Randomization occurred by assignment to either Cell 1 or Cell 2 using a randomization list, prepared by Stephens prior to the start of the study. The list was first created by concatenating blocks of size of 4 subjects, 2 for Cell 1 and 2 for Cell 2. The list was then randomized by variables from 2 independent uniform distributions: one to randomize subjects within a block and one to randomized blocks. After the randomized list was created, treatment was assigned to each subject number accordingly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cell 1: Anti-aging Serum (Active Comparator): Dosage form: Anti-aging Serum
  Frequency of Dosage: two times daily. Subjects are asked to apply 2 pumps of the Anti-aging Serum.
  Study Duration: 7 days
  Interventions: Other: Anti-aging Serum; Other: Cleansing Lotion; Other: Sunscreen
- Cell 2: Anti-aging Serum and Facial Moisturizer (Active Comparator): Dosage form: Anti-aging Serum and Facial Moisturizer
  Frequency of Dosage: two times daily. Subjects are asked to apply 2 pumps of the Anti-aging Serum, and then 2 pumps of the Facial Moisturizer to the global face.
  Study Duration: 7 days
  Interventions: Other: Anti-aging Serum; Other: Facial Moisturizer; Other: Cleansing Lotion; Other: Sunscreen

INTERVENTIONS:
Other: Anti-aging Serum — Serum composed of a patent-pending botanical extract, bioavailable peptides, antioxidants, post-biotics, and short and long-term moisturizers
Other: Facial Moisturizer — Anti-aging facial moisturizer to be used by study participants after serum
  Arms: Cell 2: Anti-aging Serum and Facial Moisturizer
Other: Cleansing Lotion — Facial cleansing lotion to be used by study participants
  Other Names: Revision Skincare® Cleansing Lotion
Other: Sunscreen — Sunscreen to be applied after application of serum in the morning. Participants were asked to reapply every 2 hours
  Other Names: Aveeno Positively Mineral Sensitive Skin SPF 40+
  Arms: Cell 1: Anti-aging Serum
Other: Sunscreen — Sunscreen to be applied after application of facial moisturizer in the morning. Participants were asked to reapply every 2 hours
  Other Names: Aveeno Positively Mineral Sensitive Skin SPF 40+
  Arms: Cell 2: Anti-aging Serum and Facial Moisturizer

SUMMARY:
This double-blind, randomized, controlled, single-center clinical trial was conducted to assess the efficacy and tolerance of an anti-aging serum to improve moderate overall photodamage and skin fatigue of aging skin after 7 days of twice-daily use when compared to the efficacy of a combination of anti-aging serum and an anti-aging facial moisturizer. A total of 26 female subjects, aged 34-60, completed study participation.

DETAILED DESCRIPTION:
This double-blind, randomized, controlled, single-center clinical trial was conducted to assess the efficacy and tolerance of an anti-aging serum (Cell 1) to improve moderate overall photodamage and skin fatigue of aging skin after 7 days of twice-daily use when compared to the efficacy of a combination of anti-aging serum and an anti-aging facial moisturizer (Cell 2). Skin fatigue was characterized by dehydrated skin with a lack of firmness (visual) and a dull appearance on the global face.

Efficacy and tolerability were assessed through clinical grading at baseline, day 3, and day 7. Efficacy evaluation on fine lines and wrinkles in the crow's feet area; overall eye appearance on the periocular area; and smoothness (tactile), firmness (visual), radiance, and overall photodamage on the global face were performed 15 minutes post product application. Self-assessment questionnaires, Glossymeter measurements, and VISIA photography were completed at baseline, day 3, and day 7.

A total of 26 subjects completed study participation, which included 12 subjects in Cell 1, and 14 subjects in Cell 2.

ELIGIBILITY:
Inclusion Criteria:

* Female, 30 to 60 years of age
* Fitzpatrick skin type I -IV
* Moderate overall photodamage of the skin
* Moderate lack of firmness (visual) of the skin
* Moderate dull appearance of the skin
* Subjects must be willing to withhold all facial treatments during the course of the study and have not undergone a treatment within the last 6 months
* Subject must be willing to provide verbal understanding and written informed consent

Exclusion Criteria:

* Diagnosed with known allergies to facial skincare products
* Nursing, pregnant, or planning to become during the duration of the study
* History of skin cancer within the past 5 years
* Having used oral isotretinoin within the last 12 months
* Having used prescription-strength skin-lightening products within the last 3 months
* Having used any anti-wrinkle, skin-lightening, or other product or topical or systemic medication known to affect skin aging or dyschromia within the last 4 weeks
* Having a health condition and/or pre-existing or dermatologic disorder that, in the Investigator's opinion, may interfere with the outcome of the study
* Having observable sunburn, suntan, scars, excessive facial hair, or other dermal conditions on the face that, in the Investigator's opinion, may influence test results
* Having a history of immunosuppression/immune deficiency disorders, or currently using oral or systemic immunosuppressive medications and biologics, and/or undergoing radiation or chemotherapy
* Using or having regularly used systemic or topical corticosteroids within the past 4 weeks
* Having started a long-term medication within the last 2 months

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Clinical Grading of Efficacy Parameters | 7 days
  The primary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10-point Scale. A decrease in scores at Day 3, and Day 7 in comparison to baseline indicates an improvement for the indicated parameter. The efficacy parameters will be assessed globally on each subject's face using a modified Griffiths' 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition):
  0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate;7 to 9 = severe (worst possible condition). The lower the score equates to the best possible outcome.
Tolerability Evaluations | 7 days
  The primary tolerability endpoint will be the Investigator Tolerability Assessment of Erythema, Edema and Dryness. A decrease in scores or lack of significant increase at Day 3, and Day 7 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example for Erythema: Erythema 0 = None No erythema of the treatment area
  1. = Mild Slight, but definite redness of the treatment area
  2. = Moderate Definite redness of the treatment area
  3. = Severe Marked redness of the treatment area

SECONDARY OUTCOMES:
Irritation Evaluation | 7 days
  The secondary tolerability endpoint will be the Subject Tolerability Assessment of Burning, Itching and Stinging. A decrease in scores or lack of significant increase at Day 3, and Day 7 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example Burning. 0 = None No burning of the treatment area
  1. = Mild Slight burning sensation of the treatment area; not really bothersome
  2. = Moderate Definite warm, burning of the treatment area that is somewhat bothersome.
  3. = Severe Hot burning sensation of the treatment area that causes definite discomfort and may interrupt daily activities and/or sleep
Self-assessment Questionnaire | 7 days
  The secondary efficacy endpoints will be the Self-Assessment Questionnaire and the Subject Treatment Satisfaction and Ease of Use Questionnaire. A decrease or increase in response values at Day 3, and Day 7 indicates an improvement compared to baseline response values. Subjects are asked to rate based on a scoring system of the following: from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement/ question being asked.
Bioinstrumentation Measurements | 7 days
  The secondary efficacy endpoints will be the Glossymeter measurements. Measurements of the gloss of the skin, taken at Day 3 and Day 7 in comparison to baseline, will measure the white light, created by LEDs, directly reflected from the skin.
VISIA-CR Photography | 7 days
  VISIA-CR photography taken at Baseline, Day 3 and Day 7 with image analysis at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Emmerich, PhD, Principal Investigator — SGS Stephens, Inc
Locations (1):
- SGS Stephens, Inc., Richardson, Texas, United States